CLINICAL TRIAL: NCT00786903
Title: Candida Spp. in the Lower Respiratory Tract: Harmless Residents or Pathogen?
Status: Completed | Type: Observational
Sponsor: Robert Krause, MD (Other)
Responsible Party: Sponsor-Investigator, Robert Krause, MD, Head, Section of Infectious Diseases and Tropical Medicine, Department of Internal Medicine, Medical University of Graz, Medical University of Graz
Organization: Medical University of Graz (Other)
Other Study IDs: 19-322 ex 07/08
Record Dates: First submitted 2008-11-05; First posted 2008-11-06 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Pulmonary Candidiasis; Invasive Candidiasis
MeSH Terms: conditions — Candidiasis, Invasive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Respiratory secretions, blood, lung tissue
Oversight: Data Monitoring Committee: Yes

SUMMARY:
In critically ill patients Candida spp. are frequently isolated from respiratory tract secretions such as endotracheal aspirates and bronchoalveolar lavages (BAL) and are most often considered as colonizers of the respiratory tract. In contrast, pneumonia due to infection with Candida spp. is rare and is diagnosed by histological demonstration of the yeast in lung tissue with associated inflammation. In spite of this, preemptive antifungal therapy based on isolation of Candida spp. from the respiratory tract is often initiated in critically ill patients. The disadvantages of this approach include increased selective pressure for the development of antimicrobial resistance, potential risks of adverse drug reactions and high treatment costs. On the other hand, immediate administration of appropriate antifungal therapy has been shown to be an important predictor of favorable outcome for patients with invasive fungal infections. Therefore, the development of reliable diagnostic measures for the detection of invasive pulmonary candidiasis is crucial. The overall objective of the proposed research project is to identify diagnostic strategies to differentiate between Candida colonization and Candida infection of the lower respiratory tract in critically ill patients. The proposed projects intends to test the hypothesis that 1.) invasive Candida strains from the lower respiratory tract differ from colonizing Candida strains with regard to production and expression of putative virulence factors and/or that 2.) patients suffering from pulmonary invasive candidiasis differ from patients colonized by Candida spp. with regard to inflammatory markers, other serum markers (fungal antigen) and composition of indigenous pulmonary bacterial flora.

DETAILED DESCRIPTION:
In critically ill patients Candida spp. are frequently isolated from respiratory tract secretions such as endotracheal aspirates and bronchoalveolar lavages (BAL) and are most often considered as colonizers of the respiratory tract. In contrast, pneumonia due to infection with Candida spp. is rare and is diagnosed by histological demonstration of the yeast in lung tissue with associated inflammation. In spite of this, preemptive antifungal therapy based on isolation of Candida spp. from the respiratory tract is often initiated in critically ill patients. The disadvantages of this approach include increased selective pressure for the development of antimicrobial resistance, potential risks of adverse drug reactions and high treatment costs. On the other hand, immediate administration of appropriate antifungal therapy has been shown to be an important predictor of favorable outcome for patients with invasive fungal infections. Therefore, the development of reliable diagnostic measures for the detection of invasive pulmonary candidiasis is crucial. The overall objective of the proposed research project is to identify diagnostic strategies to differentiate between Candida colonization and Candida infection of the lower respiratory tract in critically ill patients. The proposed projects intends to test the hypothesis that 1.) invasive Candida strains from the lower respiratory tract differ from colonizing Candida strains with regard to production and expression of putative virulence factors and/or that 2.) patients suffering from pulmonary invasive candidiasis differ from patients colonized by Candida spp. with regard to inflammatory markers, other serum markers (fungal antigen) and composition of indigenous pulmonary bacterial flora. For this purpose, pathogen related factors such as Candida prevalence, Candida quantity, phospholipases, secreted aspartyl proteinases, chromosome length polymorphism, transcriptional profiles, DFG16, SAP1-3, and SAP5 mRNA as well as human cellular and serum markers such as Dectin-1, TLR-2, TLR-4, TNF-α, IL-2, IL-10, IL-12, procalcitonin and (1→3) ß-D-Glucan, the indigenous pulmonary bacterial flora and underlying risk factors will be investigated in 6 different patient groups in this project. The results of this study should contribute to a better understanding of Candida colonization and Candida infections in the lower respiratory tract in critically ill patients. This should prospectively lead to a more targeted antifungal therapy and to a better outcome as well as to a reduction of unnecessary antifungal treatments and to a reduction of treatment costs in the future.

ELIGIBILITY:
Inclusion Criteria:

* depending on study group; i.e. no pathology of the lungs in group 1, and 4; underlying disease of the lungs in group 2 (i.e. sarcoidosis etc), infiltration of the lungs in group 3,4,5

Exclusion Criteria:

* depending on study group: i.e. HIV, recent antifungal therapy, age below 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients with and without infiltration of the lungs and with and without intubation and mechanically ventilation
Sampling Method: Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2008-11; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
pathogenic relevance of Candida in lower respiratory tract | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Robert Krause, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Styria, Austria

REFERENCES:
- [Derived] Krause R, Zollner-Schwetz I, Salzer HJ, Valentin T, Rabensteiner J, Pruller F, Raggam R, Meinitzer A, Prattes J, Rinner B, Strohmaier H, Quehenberger F, Strunk D, Heidrich K, Buzina W, Hoenigl M. Elevated levels of interleukin 17A and kynurenine in candidemic patients, compared with levels in noncandidemic patients in the intensive care unit and those in healthy controls. J Infect Dis. 2015 Feb 1;211(3):445-51. doi: 10.1093/infdis/jiu468. Epub 2014 Aug 22. PMID 25149761
- [Derived] Pruller F, Wagner J, Raggam RB, Hoenigl M, Kessler HH, Truschnig-Wilders M, Krause R. Automation of serum (1-->3)-beta-D-glucan testing allows reliable and rapid discrimination of patients with and without candidemia. Med Mycol. 2014 Jul;52(5):455-61. doi: 10.1093/mmy/myu023. Epub 2014 Jun 6. PMID 24906361